CLINICAL TRIAL: NCT03980535
Title: Evaluation of New Magnetic Resonance (MR) Imaging and Spectroscopy Software
Brief Title: New Magnetic Resonance Imaging and Spectroscopy Software in the Improvement of Image Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2011-0542; NCI-2019-02654 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0542 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device Feasibility (MRI, MRSI) (Experimental): Patients undergo an additional investigational MRI or MRSI sequence along with the standard MRI or MRSI. Healthy volunteers undergo an investigational MRI or MRSI sequence. Healthy volunteers may also undergo an additional standard sequence if there is one that can be compared to the investigational sequence. All MRI or MRSI procedures, including the standard MRI or MRSI, are no longer than 60 minutes.
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This trial studies how well new magnetic resonance imaging (MRI) and magnetic resonance spectroscopic imaging (MRSI) software works in improving the image quality of scans in both patients and healthy volunteers. Improving the image quality of MRI and MRSI through new software may lead to implementation of these techniques and better clinical care for patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To help develop and/or optimize new magnetic resonance (MR) imaging and spectroscopy applications and analysis software in order to provide the best MR services for our patients.

OUTLINE:

Patients undergo an additional investigational MRI or MRSI sequence along with the standard MRI or MRSI. Healthy volunteers undergo an investigational MRI or MRSI sequence. Healthy volunteers may also undergo an additional standard sequence if there is one that can be compared to the investigational sequence. All MRI or MRSI procedures, including the standard MRI or MRSI, are no longer than 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for routine MR imaging or spectroscopy examinations at MD Anderson Cancer Center (MDACC).
* Written informed consent will be obtained from each subject scanned who enrolled to individual sub-project under this protocol.
* HEALTHY VOLUNTEERS: Written informed consent will be obtained from each subject scanned who enrolled to individual sub-project under this protocol

Exclusion Criteria:

* No pregnant subjects will be enrolled
* No one under 18 years of age will be enrolled
* No investigational devices or drugs will be used.
* No contraindications to MR exam(s)
* HEALTHY VOLUNTEERS: No pregnant subjects will be enrolled
* HEALTHY VOLUNTEERS: No one under 18 years of age will be enrolled
* HEALTHY VOLUNTEERS: No investigational devices or drugs will be used
* HEALTHY VOLUNTEERS: No contraindications to MR exam(s) - healthy volunteers will use the same screening process utilized for MDACC patients (DI Patient Record - Part I, MR Screening Section)
* HEALTHY VOLUNTEERS: Healthy volunteers (including healthy MD Anderson employee volunteers) under the direct report of a sub-project principal investigator (PI) will be excluded for that specific sub-project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Development and/or optimization of new magnetic resonance (MR) imaging and spectroscopy applications and analysis software | Up to 7 years
  A set of images will be collected using the new magnetic resonance imaging (MRI) or MR spectroscopy techniques. Whenever appropriate, another set of images using the standard of care software will also be collected and this set of images by the standard of care software will be compared to the images that are collected with the new MRI or MR spectroscopy techniques.

CONTACTS AND LOCATIONS:
Overall Officials: John Madewell, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Saleh M, Virarkar M, Javadi S, Mathew M, Vulasala SSR, Son JB, Sun J, Bayram E, Wang X, Ma J, Szklaruk J, Bhosale P. A Feasibility Study on Deep Learning Reconstruction to Improve Image Quality With PROPELLER Acquisition in the Setting of T2-Weighted Gynecologic Pelvic Magnetic Resonance Imaging. J Comput Assist Tomogr. 2023 Sep-Oct 01;47(5):721-728. doi: 10.1097/RCT.0000000000001491. Epub 2023 Jun 9. PMID 37707401